CLINICAL TRIAL: NCT05540782
Title: Prostate Cancer Survivorship and Cognitive Health (PRO-HEALTH)
Brief Title: A Study of Cognitive Health in Survivors of Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-223
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Survivorship
Keywords: Cognitive health; Quality of Life; 22-223
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survivors of Prostate Cancer: This is a cross-sectional study with a one-time data collection process and no subsequent follow-ups. If patients did not opt out of receiving study-specific text communications, they may also receive text messages with reminders about surveys and/or direct links to REDCap to complete the surveys. Text-based communications will be delivered using the secure, HIPAA-compliant Mosio texting platform developed for clinical research.
  Interventions: Behavioral: PROMIS-SF v2.0 -Cognitive Function 8a

INTERVENTIONS:
Behavioral: PROMIS-SF v2.0 -Cognitive Function 8a — Patient-Reported Outcomes (PROs)

SUMMARY:
The purpose of this study is to collect information that may help the researchers understand the relationship between prostate cancer survivors' experiences of cancer-related cognitive dysfunction (CRCD) and their other conditions (co-morbid factors), including anxiety, depression, and insomnia. The researchers will also find out how additional things may contribute to CRCD, including social factors, the characteristics of participants' prostate cancer, and the type of cancer treatment or other medications they received.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 18 years or older
* History of histologically documented PC of any stage
* No evidence of PC Disease

Exclusion Criteria:

* <1 month since completion of surgery, radiation, chemotherapy, or ADT
* Diagnosis of Alzheimer's disease, vascular dementia, Parkinson disease, or other organic brain disorder
* Score >10 indicative of dementia on Blessed Orientation Memory Concentration

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Study Population: Patients from Memorial Sloan Kettering Cancer Center (MSK) and the Ralph Lauren Center (RLC), an MSK-affiliated Harlem community clinic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
number of participants with co-morbid symptoms | 1 year
  All participants will be evaluable as long as they have completed the PROMIS-SF v2.0 - Cognitive Function 8a.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Liou, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT05540782/ICF_000.pdf